CLINICAL TRIAL: NCT01388790
Title: Open-label, Single-arm, Multicenter Phase II Trial Investigating Cetuximab in Combination With S-1 and Cisplatin as First-line Treatment for Patients With Advanced Gastric Adenocarcinoma Including Adenocarcinoma of the Gastroesophageal Junction
Brief Title: Cetuximab in Combination With S-1 and Cisplatin in Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 062202-058
Record Dates: First submitted 2011-06-24; First posted 2011-07-07 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-09

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Cetuximab; EMD271786; TS-1; Cisplatin
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cetuximab; Cisplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab plus cisplatin plus S-1 (Experimental)
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: S-1

INTERVENTIONS:
Drug: Cetuximab — Single first dose of cetuximab 400 milligram per square meter (mg/m^2) will be administered intravenously followed by once weekly subsequent intravenous infusion of cetuximab 250 mg/m^2 in each 5-week treatment cycle until disease progression, unacceptable toxicity, or withdrawal of consent.
Drug: Cisplatin — Cisplatin 60 mg/m^2 will administered as intravenous infusion on Day 8 of each 5-week cycle maximum up to 8 cycles until disease progression, unacceptable toxicity, or withdrawal of consent
Drug: S-1 — S-1, a combination of tegafur, gimeracil, and oteracil will be administered intravenously at a dose of 40 to 60 mg/m^2 orally twice daily for first three consecutive weeks of 5-week cycle until disease progression, unacceptable toxicity, or withdrawal of consent.

SUMMARY:
This open-label, single-arm, multicenter, Phase 2 trial will treat at least 40 participants with advanced gastric adenocarcinoma including adenocarcinoma of the gastroesophageal junction (GEJ) who have not previously received systemic chemotherapy for this setting.

All eligible participants will receive the combination of cetuximab plus S-1 (a combination of tegafur, gimeracil, and oteracil) and cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and agreement with medically accepted contraception (in participants with conception potential) are obtained
* Japanese participants aged greater than or equal to 20 years
* Histologically confirmed adenocarcinoma of the stomach or GEJ (adenocarcinomas of the esophagogastric junction types I to III according to Siewert's classification) in Stage M0 (unresectable advanced) or Stage M1 (unresectable metastatic) of the disease
* Archived tumor material sample for at least subsequent standardized epidermal growth factor receptor (EGFR) expression and Kirsten-rat sarcoma (KRAS) mutation assessments
* At least one radiographically documented measurable lesion in a previously non-irradiated area according to the RECIST v 1.0
* Eastern Cooperative Oncology Group - performance status (ECOG-PS) 0 to 1
* Estimated life expectancy greater than 12 weeks
* Renal, liver and hematopoietic function as defined in the protocol.
* Sodium and potassium within normal limits or as defined in the protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Prior therapies: prior treatment with an antibody or molecule targeting EGFR- and/or vascular endothelial growth factor (VEGF) receptor-related signaling pathways; chemotherapies; or radiotherapies, major surgeries, and any investigational drugs in the 30 days before the start of trial treatment
* Concurrent chronic systemic immune or hormone therapy not indicated in this trial protocol any contraindication to treatment with cetuximab and cisplatin, or any treatments with prohibited concomitant drugs
* Brain metastasis and/or leptomeningeal disease
* Clinically relevant coronary artery disease (New York Heart Association [NYHA] functional angina classification III/IV), congestive heart failure (NYHA III/IV), clinically relevant cardiomyopathy, history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia
* Chronic diarrhea or short bowel syndrome
* Known Human Immunodeficiency Virus (HIV) infection, active or chronic carrier of hepatitis B virus (HBV) (HBV antigen positive or HBV deoxyribonucleic acid (DNA) positive) or hepatitis C virus (HCV) (HCV antibody positive)
* Pregnancy or lactation period
* Concurrent treatment with a non-permitted drug (any other chemotherapy, systemic anticancer therapy or immunotherapy)
* Previous malignancy other than gastric cancer in the last 5 years Medical or psychological conditions that would not permit the participant to complete the trial or sign the Informed Consent Form (ICF)
* Legal incapacity or limited legal capacity
* Other protocol defined exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masataka Ota, MD, Study Director — Merck Serono Co., Ltd., Japan
Locations (1):
- Please contact the Merck KGaA Communication Center located in, Darmstadt, Germany

REFERENCES:
- [Derived] Yamaguchi K, Fuse N, Komatsu Y, Fujii H, Hironaka S, Omuro Y, Muro K, Yasui H, Ueda S, Nishina T, Watanabe M, Ohtsu A. Phase II study of cetuximab plus S-1/cisplatin therapy in Japanese patients with advanced gastric cancer. Jpn J Clin Oncol. 2021 May 28;51(6):879-885. doi: 10.1093/jjco/hyaa276. PMID 33561262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): 29 June 2011/16 January 2012; Clinical data cut-off: 14 August 2012; Study completion: 13 May 2013.
Pre-assignment Details: Enrolled: 41 screened for eligibility; 1 excluded (non-fulfillment of inclusion or exclusion criteria) and 40 participants included in the study.
Groups:
- Cetuximab Plus Cisplatin Plus S-1: Cetuximab once weekly (initial dose 400 milligram per square meter [mg/m^2] followed by subsequent 250 mg/m^2 intravenous infusion), cisplatin (60 mg/m^2 intravenous infusion on Day 8 of 5-week cycle maximum up to 8 cycles) and S-1, a combination of tegafur, gimeracil, and oteracil (40 to 60 mg/m^2 orally twice daily for first three consecutive weeks of 5-week cycle) was administered until disease progression, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | Cetuximab Plus Cisplatin Plus S-1
Started | 40
Completed | 32
Not Completed | 8
Not completed — Ongoing at data cut-off date | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of study treatment.
Arm/Group | Cetuximab Plus Cisplatin Plus S-1
Number analyzed (Participants) | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR) Rate - Independent Review Committee (IRC) Assessments
Description: The best overall response rate is defined as the percentage of participants having achieved confirmed complete response plus partial response as the best overall response according to radiological assessments (based on Response Evaluation Criteria in Solid Tumors version 1.0 [RECIST v 1.0] criteria).
Time Frame: Evaluations were performed every 6 weeks until disease progression, reported between day of first participant treated, that is July 2011, until cut-off date, (14 August 2012)
Population: ITT population included all participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus Cisplatin Plus S-1
Number analyzed (Participants) | 40
percentage of participants | 40 [24.9 to 56.7]

2. Secondary Outcome: Median Progression-free Survival (PFS) Time - Independent Review Committee (IRC) Assessments
Description: The PFS time is defined as the duration from start of treatment until radiological progression (based on RECIST v 1.0 criteria) or death due to any cause within 60 days of the last tumor assessment or start of treatment. Participants without event are censored on the date of last tumor assessment.
Time Frame: Time from start of treatment to disease progression, death or last tumor assessment, reported between day of first participant treated, that is July 2011, until cut-off date, (14 August 2012)
Population: ITT population included all participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Cisplatin Plus S-1
Number analyzed (Participants) | 40
months | 5.6 [4.2 to 8.3]

ADVERSE EVENTS:
Time Frame: Time from first dose up to 30 days after the last dose of study treatment or clinical cut-off date (14 August 2012) or date of death whichever is earlier.
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to Baseline during a clinical study with an investigational medicinal product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Cetuximab Plus Cisplatin Plus S-1
Serious Adverse Events (participants affected / at risk) | 15/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Cisplatin Plus S-1 (N=40)
Acute myocardial infarction (Cardiac disorders) | 1
Pyrexia (General disorders) | 2
Electrocardiogram T wave inversion (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 6
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Renal artery thrombosis (Renal and urinary disorders) | 1
Embolism (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Trousseau's syndrome (Vascular disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Neutropenic infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hydronephrosis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Cisplatin Plus S-1 (N=40)
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 2
Trichomegaly (Congenital, familial and genetic disorders) | 2
Lacrimation increased (Eye disorders) | 5
Stomatitis (Gastrointestinal disorders) | 26
Constipation (Gastrointestinal disorders) | 25
Diarrhoea (Gastrointestinal disorders) | 24
Nausea (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 6
Cheilitis (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 19
Oedema peripheral (General disorders) | 11
Pyrexia (General disorders) | 10
Influenza like illness (General disorders) | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Paronychia (Infections and infestations) | 21
Infection (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 3
Folliculitis (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 4
Laceration (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 2
Weight decreased (Investigations) | 17
Neutrophil count decreased (Investigations) | 10
Haemoglobin decreased (Investigations) | 9
Blood creatinine increased (Investigations) | 7
Weight increased (Investigations) | 7
White blood cell count decreased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 6
Blood lactate dehydrogenase increased (Investigations) | 6
Platelet count decreased (Investigations) | 6
Protein total decreased (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 5
Blood urea increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
White blood cell count increased (Investigations) | 3
Blood amylase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood chloride decreased (Investigations) | 2
Blood urine present (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 26
Hypomagnesaemia (Metabolism and nutrition disorders) | 13
Hyponatraemia (Metabolism and nutrition disorders) | 12
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hypochloraemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dysgeusia (Nervous system disorders) | 12
Dizziness (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 30
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 21
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 12
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 11
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 7
Skin fissures (Skin and subcutaneous tissue disorders) | 7
Acne (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Skin erosion (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less